CLINICAL TRIAL: NCT06710535
Title: Global Changes Associated With Sacroiliac Joint Dysfunction and Its Reversal by Manipulation - A Randomized Controlled Trial
Brief Title: Sacroiliac Joint Dysfunction Consequences and Its Reversal by Manipulation
Acronym: LOUIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Luís Filipe Albuquerque, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aveiro University
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: Sacroiliac Dysfunction
Keywords: pain; single-leg static balance; Gait assessment; sacroiliac joint manipulation
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual manipulation (Experimental): Experimental group, subject to manipulation performed by the same Physiotherapist, using the techniques described by Shadmehr, A. et al (2018).
  Interventions: Other: Manual Manipulation
- Sham Manipulation (Sham Comparator): Sham group, subjected only to a simulation of manipulation, using the same gestures, but without manipulating, used as a placebo group.
  Interventions: Other: Sham Manipulation
- Control Group (No Intervention): Control group, which will not be subject to any intervention.

INTERVENTIONS:
Other: Manual Manipulation — The participants will receive one session of manipulation if in the experimental group. It should be mentioned that the technique will be carried out by a physiotherapist with a history of more than 10 years of manual therapy. For instance, to correct right anterior innominate rotation, the participant will be made to lie on the side so that the affected side is upward. The physiotherapist will stand in front of the participant; first we will put their shoulders, pelvis and lower limbs in neutral position and place the right hand on the anterior superior iliac spine (ASIS) and the left hand on the ischium tuberosity and with a rotational movement of the hands, the physiotherapist will rotate the ilium posteriorly. At the end of the range, we will replace the position of hands and place the left forearm on the ischium tuberosity and place the right hand on the upper participant's shoulder and will move it toward the bed at the end of the range in exhalation a thrust will be executed.
  Arms: Manual manipulation
Other: Sham Manipulation — The participants will receive one session of sham manipulation if in the sham group. For instance, to correct right anterior innominate rotation, the participant will be made to lie on the side so that the affected side is upward. The physiotherapist will stand in front of the participant; first we will put their shoulders, pelvis and lower limbs in neutral position and place the right hand on the anterior superior iliac spine (ASIS) and the left hand on the ischium tuberosity and with a rotational movement of the hands, the physiotherapist will rotate the ilium posteriorly. At the end of the range, we will replace the position of hands and place the left forearm on the ischium tuberosity and place the right hand on the upper participant's shoulder and will move it toward the bed at the end of the range in exhalation, the physiotherapist will pretend to execute a thrust.
  Arms: Sham Manipulation

SUMMARY:
Sacroiliac joint dysfunction (ASI) is an alteration in the normal biomechanics of the joint, which leads to hypomobility or hypermobility of that joint. It is one of the most common causes of misdiagnosis in low back pain and when not treated correctly, it often evolves into chronic pain (30% to 42%) and disability. Manipulating the dysfunctional ASI appears to result in benefits and significantly positive changes at various levels, in all segments of the human body. With this investigation, the investigators intend to clarify and deepen the possible correlation between the changes that normally accompany this dysfunction, as well as its possible reversibility with its normalization.- Objectives

* The investigators will essentially have two main objectives:

  1. Mapping of the most evident symptomatic changes, when sacroiliac joint dysfunction is present, in terms of pain, balance and gait ;
  2. To try to understand the immediate, global and short-term effect of ASI manipulation, studying the cumulative effect of six sessions and the possible interrelationship between the changes recorded.

     - Study design Quantitative, with experimental study design, RCT, with the sample comprising individuals with SIJ dysfunction, where all participants in study 2 will be randomly allocated to the experimental, control and placebo groups. It will be carried out at the University of Aveiro facilities.

     Initially, the investigators will map the changes present at a physical level, followed by manipulation, evaluating the immediate effect, measuring the degree of pain, unipodal balance and satisfaction with the treatment.

     The investigators will then evaluate the effect of 3 sessions, on a weekly basis, for 3 weeks.

     - Material and methods

     The investigators will make use of:
* Standing flexion test, to define the laterality of the dysfunction;
* VAS , to subjectively assess pain;
* Pressure algometer, to objectively assess pain ;
* Force Platform, to assess balance;
* G-Walk, for gait assessment;
* PGIC, to assess satisfaction with treatment ;

DETAILED DESCRIPTION:
Procedures to be used in the Experimental Study Material and methods

Reception of participants, with a clear explanation of the objectives and procedures to be used in the pilot study, asking them to fill out:

1. an informed consent model; 2. a sociodemographic and health data questionnaire; 3. a participant recruitment form (all of which were previously approved by the Data Protection Officer and the Ethics and Deontology Council of the University of Aveiro); 4. Select the study participants, assessing the presence of Sacroiliac Joint Dysfunction, for which the investigators will use the following procedures, using a multitest assessment, which consists of using a combination of palpation and pain provocation tests, which exhibits sufficient validity and reliability in the diagnosis of sacroiliac joint dysfunction ( Telli et al., 2018); 4. 1 - Bending test in foot - Performed by palpating the posterior superior iliac spine (PSIS) while the person is bending forward from the standing position. The test is negative if PSISs appear to move equally and sym - metrically, or positive on the side in which the PSIS moves crani - ally and ventrally more than the other side. A positive result indicates limited movement of the ilium on the sacrum, and therefore limited SIJ movement on the side of the superior PSIS ( Ribeiro et al, 2021); 4.2 - Bending test sitting - Similar to the standing flexion test, but the persons starts from the sitting position. The test is negative if PSISs appear to move equally and symmetrically, and positive on the side on which the PSIS moves cranially and ventrally more than the other side. A positive result indicates limited movement of the sacrum on the ilium, and therefore limited SIJ movement on the side of the superior PSIS (Ribeiro et al, 2021); 4.3 - Thigh thrust test (POSH) - The patient lies in a supine position. The hip is brought to 90º flexion. Pressure is applied directly toward the examination table. Pathology in the SI joint is considered if pain occurs in the hip. Pain provocation is established with hip flexion and adduction ( Telli et al, 2018); 4.4 - Sacral thrust test - The patient lies in a prone position. The practitioner places one hand on the apex of the sacrum while applying direct pressure with the other hand ( Telli et al, 2018); 4.5 - FABER test - The patient lies in a supine position, while the practitioner stands beside the patient and bends the patient's knee, bringing the heel to the opposite knee. With the other hand, the investigator ensures that the contralateral anterior superior iliac spine remains in a neutral position. The doctor applies mild pressure to the bent knee. Pressure is assumed to be applied to the bilateral sacroiliac ligaments and hip joints. Pain provocation occurs with flexion, abduction and external rotation of the hip ( Telli et al, 2018)

Participants who test positive in at least 4 of the 5 tests mentioned above will be selected to participate in the following studies:

- PHASE 1 Objective : mapping of changes present in selected individuals with SIJ dysfunction, in terms of pain, unipedal static balance and gait;

Variables :

* Pain;
* Static balance;
* Single-leg static balance;
* Gait assessment;

Instruments : -

* Visual Analogue Scale (VAS) , to assess the subjective sensation of pain perceived by the participant;
* Pressure Algometer , to assess pain, used at the following points:

  * Lower limbs: muscular belly of the external calves, 8 cm below their origin and muscular belly of the internal calves, 12 cm below the origin, cuboids and tarsal naviculars, external and internal joint interline, middle third, in both knees
  * Upper limbs: bilaterally at the level of the muscular belly of the short portion of the biceps brachii, 9 cm above the elbow crease and muscular belly of the long portion of the same muscle, 9 cm above the elbow crease , epicondyle and epitrochlea.
  * Cervical spine: At the level of the transverse processes of C4, bilaterally;
  * Lumbar spine: At the level of the transverse processes of L3, bilaterally;
  * Sacroiliac joints bilaterally, at the level of the posterior superior iliac spine, bilaterally;
  * Craniocervical transition, bilaterally, at the level of the occipital origin of the upper trapezius muscle;
* Force platform , to assess single-leg static balance;
* G-Walk, wearable inertial sensor for motion analysis, for gait assessment;

  * PHASE 2 Objective : To evaluate the immediate effect of ASI manipulation, assessing the variables at the beginning and end of the first session, regarding pain, balance, gait assessment, overall perception of change and satisfaction with the intervention, with weekly frequency, for 3 weeks.

Clinical trial (RCT), in which participants will be randomly divided into 3 groups:

1. Experimental group , subject to manipulation performed by the same Physiotherapist, using the techniques described by Shadmehr, A. et al (2018);
2. Sham Group , subjected only to a simulation of manipulation, using the same gestures, but without manipulating, used as a placebo group;
3. Control group , which will not be subject to any intervention.

Variables :

* Pain;
* Single-leg static balance;
* Gait assessment;
* Perception of change and satisfaction with treatment.

Instruments:

* VAS, used before and immediately after the intervention ;
* Pressure algometer, evaluating before and immediately after the intervention ;
* Force platform;
* G-Walk, wearable inertial sensor for motion analysis, for gait assessment;
* PGIC , to assess the perception of change and satisfaction with treatment, immediately after the last treatment;

ELIGIBILITY:
Inclusion Criteria:

* Participants with sacroiliac joint dysfunction demonstrated
* Students of Aveiro University
* Aged between 18 and 30 years

Exclusion Criteria:

* Individuals with neurological injuries
* Subject to another type of therapeutic intervention, during the intervention period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Subjective Pain Assessment | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week]
  Pain will be assessed with the Visual Analogue Scale (VAS), a horizontal line graded 0 (better outcome) to 10 (worse outcome).
Algometry Pain Assessment | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week
  Pressure algometer
Single-leg balance | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week]
  Assess single-leg balance with a force platform
Gait parameters | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week
  Assess gait parameters with G-Walk, a wearable inertial sensor for motion analysis
Global perception of change and satisfaction with treatment | Immediately after the last treatment
  PGIC ( Patient Global Improvement Change Scale ) - is an instrument for measuring and evaluating the global perception of change and satisfaction with treatment, used in any health condition, unidimensional, with a scoring system on a positive orientation scale from 1 to 7, with a completion time of 1 minute*.

CONTACTS AND LOCATIONS:
Locations (1):
- Aveiro University, Aveiro, Portugal